CLINICAL TRIAL: NCT05643963
Title: modifiCatiOn of fOod intaKe to Influence the Equilibrium of the uRinary BLADDER
Brief Title: The COOKER-BLADDER Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roland Seiler-Blarer (Other)
Responsible Party: Sponsor-Investigator, Roland Seiler-Blarer, Prof. Dr. med., Hospital Centre Biel/Bienne
Organization: Hospital Centre Biel/Bienne (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: SZB-URO-23-001
Record Dates: First submitted 2022-11-04; First posted 2022-12-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Diet, Healthy; Urinary Bladder Diseases; Oncogenesis
MeSH Terms: conditions — Urinary Bladder Diseases; Carcinogenesis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focus on bladder protective diet (Experimental): For 12 weeks, healthy volunteers will follow a bladder protective diet.
  Interventions: Other: Dietary regimens
- No focus on bladder protective diet (Experimental): For 12 weeks, healthy volunteers will not follow a specific diet.
  Interventions: Other: Dietary regimens

INTERVENTIONS:
Other: Dietary regimens — Food intake will follow a recommendation according to a specific list. Protective and non-protective food intake will be performed for specific time periods with biomarker assessment after each period.

SUMMARY:
The goal of this interventional study is to test the influence of food intake with characteristics of the urinary bladder. The main questions it aims to answer are:

* How does food intake modify the characteristics of urothelial cells?
* Does change of specific diet regimes influence biomarker characteristics in urine? Participants will follow specific diet regime for a given time period. After completion of this period biomarker assessment is performed. Thereafter the participants follow an opposite diet regime for the same time period with identical biomarker assessment at the end.

Biomarkers within the participants and between the diet regimes will be compared to investigate the influence of food intake on the urinary bladder.

ELIGIBILITY:
Inclusion Criteria:

* no daily medication
* no ongoing medical treatment

Exclusion Criteria:

* Chronic disease
* Regular medication
* Not willing to follow diet instructions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Change in molecular profile of urothelial cells | 12 weeks
  After the 12 week diet period (protective and non-protective), cells voided in urine will be sampled and examined.

SECONDARY OUTCOMES:
Change in multiplex cytokine levels in voided urine | 12 weeks
  After the 12 week diet period (protective and non-protective), supernatant in voided urine will be used for further examination
DNA sequences in urinary microbiome | 12 weeks
  After the 12 week diet period (protective and non-protective), DNA sequencing on urinary microbiome in voided urine will be performed and compared between the different dietary regimens.
Change of BMI | 12 weeks
  After the 12 week diet period (protective and non-protective) BMI will be assessed.
Change of heart rate | 12 weeks
  After the 12 week diet period (protective and non-protective), heart rate will be assessed.
Change of blood pressure | 12 weeks
  After the 12 week diet period (protective and non-protective), systolic and diastolic blood pressure will be assessed.
Change of health status | 12 weeks
  After the 12 week diet period (protective and non-protective), health status will be assessed using the Short Form 36 (SF-36) questionaire.
  The possible score ranges from 0 to 100 points, with 0 points representing the greatest possible health limitation, and 100 points representing no health limitation.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Department of Urology, Spitalzentrum Biel, Biel/Bienne, Canton of Bern
  - Roland Seiler, Biel

IPD SHARING:
Plan to Share IPD: Yes
Data from biomarker assessment and diet regimens will be provided in the general public
Supporting Information: Study Protocol, Analytic Code
Time Frame: At publication